CLINICAL TRIAL: NCT03685747
Title: A Prospective, Single-site, Open-label, Pharmacokinetic Study of Intermittent Intraperitoneal Vancomycin in Adult Subjects Receiving Automated Peritoneal Dialysis
Brief Title: Vancomycin Pharmacokinetics in Patients on Peritoneal Dialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Walter K. Kraft, Clinical Research Unit Medical Director, Thomas Jefferson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12451
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Peritoneal Dialysis-associated Peritonitis
Keywords: Vancomycin; Pharmacokinetics; Pharmacodynamics; Automated Peritoneal Dialysis
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vancomycin (Experimental): A single 20 mg/kg intraperitoneal dose in 1-liter of 7.5% icodextrin solution of vancomycin will be administered. Sparse blood sampling will be obtained during an overnight 12-hour dwell and during the exchange period.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Vancomycin one-time 20 mg/kg intraperitoneal dose.

SUMMARY:
Vancomycin is the most commonly used empiric treatment for infectious peritonitis in patients on peritoneal dialysis. Current dosing and monitoring for safety and efficacy is empiric, especially for those on rapid-cycling modalities. The goal of this study is to understand the pharmacokinetics of vancomycin in patients on rapid-cycling peritoneal dialysis modalities in order to derive an optimal dosing regimen.

DETAILED DESCRIPTION:
Peritoneal dialysis (PD) is a form of renal replacement therapy indicated for those with acute kidney injury or end stage renal disease. Currently, two modalities of PD exist and is individualized based on patient and life-style specific factors. Continuous ambulatory peritoneal dialysis (CAPD) allows 4 - 5 exchanges performed manually whereas automated peritoneal dialysis (APD) involves continuous, automated, cyclical exchanges performed by a device at home during the night. Peritonitis is a common complication in PD and accounts for a large portion of hospital readmission and mortality. Vancomycin is the most common antibiotic recommended and has notable gram-positive coverage used empirically during suspected peritonitis.

Despite widespread use, vancomycin lacks good pharmacokinetic characterization in PD. Early pharmacokinetic studies using vancomycin were conducted predominantly in patients on CAPD on glucose-based prescriptions. Data is non-existent in PD patients administered the novel dialysate solution icodextrin, or those treated with overnight APD. The impact of residual kidney function (RKF) on vancomycin in PD is also lacking. Enhanced vancomycin clearance in RKF may result in under-dosing, while overdosing may result in nephrotoxicity and loss of clinically important RKF.

The investigators will characterize the pharmacokinetic profile of vancomycin following a single intraperitoneal dose of vancomycin in icodextrin dialysate to non-infected PD patients and examine the relationship between RKF and vancomycin clearance using serum, dialysate and urine. The goal is to use this data in non-infected subjects to generate information to guide vancomycin dosing in patients on rapid-cycling PD modalities.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or females between 18 - 85 years old
* Stabilized on a PD regimen for > 3 months prior to study initiation

Exclusion Criteria:

* Clinically significant disease unrelated to renal impairment or deemed unfit by the investigator
* Allergy or hypersensitivity to vancomycin or icodextrin-containing dialysis solution
* Active peritonitis infection
* Previous intraperitoneal antibiotic treatment within 2 months
* Previous intravenous vancomycin treatment within 2 months
* Hemoglobin < 9 g/dL
* Pregnant or breast-feeding women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter K Kraft, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual level PK de-identified data maybe shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: through 2024
Access Criteria: email. walter.kraft@jefferson.edu

REFERENCES:
- [Result] Lam E, Ting Kayla Lien Y, Kraft WK, Stickle DF, Piraino B, Zhang J. Intraperitoneal pharmacokinetics of vancomycin in patients on automated peritoneal dialysis. Clin Transl Sci. 2022 Mar;15(3):649-657. doi: 10.1111/cts.13182. Epub 2021 Nov 9. PMID 34755479

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vancomycin
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vancomycin
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Total Plasma Concentration (Cmax)
Description: Total systemic plasma concentration following 12-hour dwell
Time Frame: Day: 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Vancomycin
Number analyzed (Participants) | 4
mg/L | 28.7 (4.9)

2. Primary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Time (hours) to achieve the maximum plasma concentration
Time Frame: Day: 1
Measure: Median (Full Range); unit: hours
Arm/Group | Vancomycin
Number analyzed (Participants) | 4
hours | 14.4 [13.8 to 15]

3. Primary Outcome: Area Under the Concentration-time Curve (AUC0-inf)
Description: AUC based on vancomycin plasma concentrations
Time Frame: Days: 1-7
Measure: Mean (Standard Deviation); unit: hr x mg/L
Arm/Group | Vancomycin
Number analyzed (Participants) | 4
hr x mg/L | 2589.9 (365.6)

4. Primary Outcome: Total Body Clearance (CLtotal)
Description: Total vancomycin plasma vancomycin clearance
Time Frame: Days: 1-7
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Vancomycin
Number analyzed (Participants) | 4
mL/min | 7.2 (1.3)

5. Primary Outcome: Dialytic Clearance
Description: Vancomycin clearance from peritoneal dialysis
Time Frame: Days: 1-7
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Vancomycin
Number analyzed (Participants) | 4
mL/min | 11.1 (4.3)

6. Secondary Outcome: Adverse Events
Description: Any adverse events throughout entirety of study as assessed by physician-investigator
Time Frame: Days: 1-7
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: 10 days
Description: Subjects were assessed daily for adverse events till day 7 and then again on day 10 post study visit
Arm/Group | Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT03685747/Prot_SAP_000.pdf